CLINICAL TRIAL: NCT03592680
Title: Influence of Oral Vitamine C Supplementation on the Incidence of Post-operative Atrial Fibrillation
Brief Title: Influence of Vitamin C on Post-operative Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Dr. Alain Kalmar, MD, PhD, Staff Anesthesist, Algemeen Ziekenhuis Maria Middelares
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MMS.2017.011
Record Dates: First submitted 2018-06-22; First posted 2018-07-19 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation
Keywords: Post-operative atrial fibrillation; Ascorbic Acid; Vitamin C; antioxidant; Cardiac surgery
MeSH Terms: conditions — Atrial Fibrillation | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: One group receives Vitamin C, the other group received placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C (Active Comparator): Vitamin C 1000mg PO from 5 days before surgery until 10 days after surgery
  Interventions: Dietary Supplement: Vitamin C
- Placebo (Placebo Comparator): Placebo as an alternative for Vitamin C tablets
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C — 1 gram Vitamin C will be administrated orally, twice a day from 5 days before until 10 days after surgery.
  Arms: Vitamin C
Other: Placebo — 1 gram Placebo will be administrated orally, twice a day, from 5 days before until 10 days after surgery
  Arms: Placebo

SUMMARY:
Post-operative atrial fibrillation (POAF) is the most common arrhythmia which typically develops 2-3 days after cardiac surgery. The incidence of POAF variates between 10% and 65% depending on the type of cardiac surgery and is especially high in patients which underwent Coronary Artery Bypass Grafting (CABG) and heart valve surgery. POAF is associated with increased morbidity and mortality and has a major impact on hospital resources.

The precise pathogenesis of POAF is very complex, but several studies have demonstrated an association between inflammation, oxidative stress and POAF. Since this oxidative stress may be reduced by dietary anti-oxidantia such as vitamin C, the aim of this study is to evaluate the effect of oral vitamin C administration of the incidence of POAF.

DETAILED DESCRIPTION:
After obtaining informed consent, patients which are planned for CABG or heart valve surgery are randomly assigned into the Vitamin C group or Placebo Group.

Each patient will receive 1 g Vitamin C or Placebo twice a day from 5 days before until 10 days after surgery. The medication will be given orally and both patient and surgeon are blinded for the administrated medication.

Patients receive standard of care in the post-operative period, which includes close monitoring for possible arrhythmias. If such an arrhythmia develops, this is treated according to the normal procedures. All information such as the used medication, the hospitalization / ICU length of stay and the ventilation time is automatically registered in the patient records.

From each patient, three additional blood samples (peri-operative, post-operative Day 0, post-operative Day 1) will be obtained for analysis of Neutrophil gelatinase-associated lipocalin (NGAL), a possible marker of subclinical kidney damage. These samples will be analysed in batch once all samples are collected.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* eligible for elective cardiac surgery
* preoperative sinus rhythm

Exclusion Criteria:

* patients who do not want to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Arrhythmia | First 5 days postoperatively
  Incidence

SECONDARY OUTCOMES:
hours of endotracheal ventilation | from arrival at ICU after surgery until the time of discharge from ICU. average 48 hours.
  number of hours of endotracheal ventilation after surgery
Length of stay at ICU | from time of arrival at ICU after surgery until the time of discharge from ICU. upto 14 days. average 48 hours.
  number of hours in the Intensive Care Unit
Length of stay in the hospital | from time of arrival at ICU after surgery until the time of hospital discharge. upto 120 days.
  number of hours in the hospital
Cost of postoperative medication | from time of arrival at ICU after surgery until the time of hospital discharge. upto 120 days
  Total cost (€) of postoperative medication
subclinical kidney damage | after induction of anesthesia and two hours after CPB
  change in Value of NGAL between pre-incision and post-CPB
Postoperative complications | from time of arrival at ICU until the time of hospital discharge. upto 120 days
  Number of unexpected complications requiring medical interventions

CONTACTS AND LOCATIONS:
Overall Officials: Alain F Kalmar, MD, PhD, MSc, Principal Investigator — Maria Middelares Hospital
Locations (1):
- AZ Maria Middelares, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Heerman J, Boydens C, Allaert S, Cathenis K, Deryckere K, Vanoverschelde H. Effect of Perioperative Oral Vitamin C Supplementation on In-Hospital Postoperative Medication Costs for Cardiac Surgery Patients: A Prospective, Single-Centre, Randomised Clinical Trial. Pharmacoecon Open. 2023 Jul;7(4):655-663. doi: 10.1007/s41669-023-00412-3. Epub 2023 Apr 11. PMID 37039967